CLINICAL TRIAL: NCT06678087
Title: The Effect of Birth and Motherhood Preparation Meditation Given with Thetahealing Meditation Method on Fear of Birth, Normal Birth Belief and Self-Efficacy and Normal Birth Rate
Brief Title: Meditation for Preparation for Birth and Motherhood Given with Thetahealing Meditation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, FatmaZehra AKPINAR, phd student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ataturk Uni.
Record Dates: First submitted 2024-10-16; First posted 2024-11-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Meditation; Fear of Labor; Thetahealing Meditation
Keywords: Brain; birth; Fear of Birth; Preparation for Birth; Pregnancy Education; EEG; Brain Waves; Meditation; Complementary and Alternative Medicine; ThetaHealing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A control group (No Intervention): This is the group that receives routine antenatal care.
- Group B Pregnancy School (Other): This is a group of pregnant women who receive birth preparation training at the hospital's pregnancy school in addition to routine antenatal care.
  Interventions: Other: pregnancy school,
- group c experimental group (Experimental): In addition to routine antenatal care and childbirth preparation training at the hospital's pregnancy school, this group will receive childbirth and motherhood preparation meditation training prepared with the thetahealing meditation method simultaneously with the childbirth preparation training.
  Interventions: Other: motherhood preparation meditation training prepared with the thetahealing meditation method

INTERVENTIONS:
Other: motherhood preparation meditation training prepared with the thetahealing meditation method — With Birth and Motherhood Preparation Meditation, all physiological and psychological reasons causing fear of birth will be addressed. How to do the meditation will be taught by the practitioner in the course.
  The root belief analysis study for each topic is carried out with the questions of who, what, when, where, why and how. Then, the reprogramming work that allows the change of that belief, feeling, emotion will be done with methods specific to the technique.
  The topics to be worked on during meditation each week are listed below. Each week, pregnant women will be given a 15-minute meditation homework per day until the next week regarding the topic worked on.
  All meditations begin with relaxation and breathing exercises. In each meditation, the emotion and root-belief analysis related to the relevant topic will be done by the practitioner.
  With this application, it is aimed to accelerate the change in the mind with positive language and regular repetition.
  Arms: group c experimental group
Other: pregnancy school, — In the pregnancy school, an informational support training is provided to pregnant women and their families to ensure that the pre-pregnancy, pregnancy and birth process is passed in a healthy and conscious manner.
  The training content includes:
  Reproductive organs and development, Nutrition during pregnancy and puerperium, Common problems during pregnancy, Physiological changes, Non-formological methods, Breathing techniques during birth, Anesthetic methods, Birth methods and techniques, Postpartum and baby care, Newborn Care / Problems, Home-Bag-Hospital preparation, Breast milk - Its importance - Breastfeeding, Family planning topics are given five days a week for 2 hours.
  Arms: Group B Pregnancy School

SUMMARY:
Fear of childbirth If left untreated, it negatively affects women's birth process and preferences. Determining the level of fear experienced by women during pregnancy and helping them cope with this fear will help reduce the negative effects.

Theta-Healing is defined as a deep meditation method based on the belief that all unwanted situations that occur in humans originate from the subconscious of the human mind and that healing will occur when the beliefs in the subconscious are resolved and changed to be beneficial to the individual.

This study aims to help women with different levels of fear of childbirth cope with fear by revealing the reasons for their subconscious fear of childbirth with the ThetaHealing meditation method.

This study, which is planned to be conducted as a randomized controlled trial design, aims to present a new method in midwifery care to be applied for the management of pathological fear of childbirth. In addition, it is aimed to reduce the fear of pathological childbirth and increase normal birth self-efficacy and increase the normal birth rate.

The study is planned as a randomized controlled experimental study. Pregnant women will be randomized in accordance with the randomization rules. For randomization, the Random Integer Generator method in the Numbers subheading of the https://www.random.org site will be used to.

The study consists of a total of 3 groups, namely the control group (A) and the experimental groups (B, C).

* Group A will be the group that receives routine hospital and midwifery care (n=30)
* Group B will be the group that receives childbirth preparation training at the hospital's pregnancy school in addition to routine care (n=30)
* Group C will be the group that receives childbirth preparation training at the hospital's pregnancy school in addition to routine care and will additionally receive a childbirth and motherhood preparation meditation created with theta-healing method (n=30).

The research will be conducted between May and December 2024 among pregnant women who apply to the Ankara City Hospital Gynecology and Obstetrics Department and agree to participate in the study.

After the groups are formed, the researcher will collect research data from all groups using a personal information form, the Fear of Childbirth Sub-Dimension Scale of the Prenatal Self-Assessment Scale, the Self-Efficacy Scale for Normal Birth, and the Normal Birth Belief Scale.

DETAILED DESCRIPTION:
The study consists of a total of 3 groups, namely the control group (A) and the experimental groups (B, C).

* Group A is the group that receives routine hospital and midwifery care,
* Group B is the group that receives birth preparation training at the hospital's pregnancy school in addition to routine care,
* Group C is the group that receives birth preparation training at the hospital's pregnancy school in addition to routine care and is additionally applied to birth and motherhood preparation meditation created with theta-healing method.

The trainings at the Ankara City Hospital Gynecology and Obstetrics Department Pregnancy School are held every weekday at 10:00 and 12:00 and continue as a weekly program.

The contact information of all participants will be collected at the beginning so that contact can be made and planning can be made in the later stages of the study.

After the groups are formed, the researcher will collect the personal information form, the Prenatal Self-Assessment Scale Fear of Birth Sub-Dimension Scale, Self-Efficacy Scale for Normal Birth and the Belief in Normal Birth Scale and pre-test data for all groups.

Then, all groups will watch a 6-minute birth video containing various birth images while simultaneously recording their brain waves with a mobile EEG device.

In the 2nd step of the study (intervention step), while Group C continues to receive birth preparation training at the pregnancy school, the birth and motherhood preparation meditation study prepared with the theta-healing meditation method will be carried out by the researcher who is a theta-healing practitioner who has received training on this subject.

At the end of the Birth Preparation Training and Meditation study given at the pregnancy school, the experimental (B, C) and control (A) groups will be shown the birth video used at the beginning of the study for 6 minutes, as in the beginning of the study, and during this time, their brain activities will be recorded for the second time with the mobile EEG device. Then, post-test data will be collected again with the Prenatal Self-Assessment Scale Fear of Birth Sub-Dimension Scale, Self-Efficacy Scale for Normal Birth and Normal Birth Belief Scale.

Later, all pregnant women included in the study will notify the researcher at the beginning of labor and their brain activity will be recorded for 6 minutes with a mobile EEG device during labor. Finally, it is aimed to determine the level of fear experienced during and after labor by using the Wijma Birth Expectation/Experience Scale (W-DEQ) between the 1st and 10th day after labor.

ELIGIBILITY:
Inclusion Criteria:

1. Being primiparous pregnant.
2. Being between the ages of 18-50.
3. Being a high school graduate.
4. Not having vision or hearing problems.
5. Not having communication problems.
6. Not having a risky pregnancy.

Exclusion Criteria:

1. Not having a high school graduate.
2. Being a multiparous pregnant woman.
3. Having a vision or hearing problem.
4. Having a communication problem.
5. Being diagnosed with a risky pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 and over, pregnant
Enrollment: 100 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prenatal Self-Assessment Scale- Fear of Birth Sub-Dimensions Description | 1st measurement: at the first meeting with all study groups 2nd measurement: group a 5 days after the 1st measurement. group b and group c at the end of the training.
  he scale is used to evaluate the adaptation of pregnant women to pregnancy and motherhood. The "Fear of Birth" subscales in the scale will be used. Items are evaluated with scores ranging from "1" to "4" (4: "Describes very much," 3: "Partly describes," 2: "Somewhat describes," 1: Does not describe at all"). The lowest score to be taken separately in the fear of birth and birth readiness sub-dimensions is 10 and the highest score is 40.
Normal Birth Belief Scale (NBS) | 1st measurement: at the first meeting with all study groups 2nd measurement: group a 5 days after the 1st measurement. group b and group c at the end of the training.
  Developed by Akça and Aksoy Derya in 2021 in line with the Health belief model, NBS evaluates the beliefs and tendencies of pregnant women regarding normal birth. The NEQ consists of 6 sub-dimensions and 24 items: perceived susceptibility (items 1, 2, 3), perceived severity (items 4, 5, 6, 7), perceived benefits (items 8, 9, 10, 11), perceived barriers (items 12, 13, 14, 15, 16, 17), perceived self-efficacy (items 18, 19, 20, 21) and health motivation (items 22, 23, 24). The items in the scale are five-point Likert-type and are scored as "I completely agree (5)", "I agree (4)", "I am undecided (3)", "I disagree (2)", "I completely disagree (1)". All items belonging to the NEQ perceived barriers sub-dimension (items 12, 13, 14, 15, 16, 17) are reverse scored. The lowest possible score is 24 and the highest possible score is 120. The lowest possible scores are 3 and 15 from the "perceived susceptibility" sub-dimension, lowest possible scores are 4 and 20 from the "perceived seriousness"
Self-Efficacy Scale for Normal Birth | 1st measurement: at the first meeting with all study groups 2nd measurement: group a 5 days after the 1st measurement. group b and group c at the end of the training.
  The scale developed by Chu et al. (2017) is a Thurstone type scale consisting of 9 items. Each item of the measurement tool is scored as "0 points = I don't trust myself, 10 points = I am very confident". The lowest score that can be obtained from the scale is 0, while the highest score is 90. As the scores obtained from the self-efficacy scale increase, the level of self-efficacy also increases. The total Cronbach Alpha value of the original scale is 0.93.
Wijma Childbirth Expectation/Experience Scale (W-DEQ) Version B | Measurement between 1-10 days after birth for all groups will be taken.
  This scale was developed by Wijma and colleagues. The aim of the scale is to assess women's fear of childbirth during their own childbirth experiences in the postpartum period. The validity and reliability study for our country was conducted by Uçar and Beji (29). The scale consists of 33 items. Each item is a 6-point Likert-type scale with scores ranging from 1 to 6, with 1 being "completely" and 6 being "not at all". The minimum score on the scale is 33, while the maximum score is 198. High scores indicate that women have high fear of childbirth. The negative loaded questions in the scale (2, 3, 6, 7, 8, 11, 12,15, 19, 20, 24, 25, 27, 31) are calculated by turning them in the opposite direction in order to ensure consistency in the measurement. W-DEQ scores are evaluated in four subgroups.
  These are; women with low-level fear of childbirth (W-DEQ score ≤37), women with moderate-level fear of childbirth (W-DEQ score between 38-65), women with severe fear of childbirth (W-DEQ score 6
Brain Wave Measurement with Mobile EEG Device | 1st measurement: at the first meeting with all study groups 2nd measurement: group a 5 days after the 1st measurement. group b and group c at the end of the training. 3rd measurement: at the time of labor for all groups.
  While all participants will watch 6-minute images of different births, their brain waves will be recorded with a mobile EEG device to record the participants' brain responses to the birth.

CONTACTS AND LOCATIONS:
Overall Officials: serap ejder apay, Principal Investigator — ATATURK UNI.
Locations (1):
- Ataturk Uni, Erzurum, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No